CLINICAL TRIAL: NCT03990090
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Phase Ia Study in Chinese Healthy Adult Subjects to Investigate the Safety, Tolerability and Pharmacokinetic of TG103
Brief Title: A Study of TG103 in Chinese Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TG103/201901
Record Dates: First submitted 2019-06-12; First posted 2019-06-18 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: TG103; Pharmacokinetic; Pharmacodynamic; Safety; Tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TG103 (Experimental): Escalating doses of TG103 administered subcutaneously (SC) once in healthy participants.
  Interventions: Drug: TG103
- Placebo (Placebo Comparator): Placebo administered SC once in healthy participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TG103 — Administered SC
  Arms: TG103
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purposes of this study are to determine:

1. To assess the safety and tolerability of a single subcutaneous injection of different doses of TG103 in healthy Chinese adult subjects.
2. The pharmacokinetic and pharmacodynamic characteristics of a single subcutaneous injection of different doses of TG103 in healthy Chinese adult subjects were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and ≤ 65 years old, male or female;
* Medical history, physical examination, vital signs, 12-lead ECG and laboratory examination, imaging examination (thyroid color Doppler ultrasound, abdominal color Doppler ultrasound, chest X-ray) in the normal range, or not in the normal range but the researchers consider they have no clinical significance;
* The weighing no less than 50 kg in male subjects, and no less than 45 kg in female subjects , body mass index (BMI) between 18.9 and 27.9 kg/m2 (including boundary values)
* Fasting blood glucose is between 3.9-6.1 mmol/L (excluding the boundary value), and HbA1c is <5.7%;
* Subjects must use reliable methods of contraception throughout the study period and avoid pregnancy in women or pregnancy in male subjects' partners at least 3 months after dosing;
* The subject is fully aware of the test content and possible adverse reactions, and has the ability to communicate properly with the researcher while complying with the research requirements;
* Voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

* Have a history of severe drug or food allergies, or who may be allergic to the test drug by the investigator;
* Have serious history of pancreas, liver, kidney, gastrointestinal tract, cardiovascular, respiratory, hematological, central nervous system disease, etc.，or other important disease that have risks may endanger the safety of the subject or affect the absorption, metabolism, excretion, etc. of the study drug，or the investigator believes that the subject is not suitable for inclusion.
* Have undergone major surgery within 3 months prior to the trial, or have experienced severe infection within 4 weeks prior to the trial;
* Have diabetes, thyroid dysfunction or other endocrine diseases that may affect blood sugar metabolism;
* Individual or family history of medullary thyroid carcinoma (MTC) or type 2 multiple endocrine neoplasia, or other genetic diseases that are susceptible to medullary medullary cancer;
* Those with history of malignant tumors and mental illness, depression, anxiety, and epilepsy disease.
* Drugs and drug abusers in the past three years;
* Vaccination within 28 days prior to the trial or planned to be vaccinated within 1 week of receiving the study drug;
* Has one or more positive tests in Hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or anti- Treponema pallidum-specific antibody;
* Lost more than 400 ml of blood due to blood donation or other reasons within 3 months before the test;
* Apply a glucagon-like peptide-1(GLP-1 )analogue, a glucagon-like peptide-1(GLP-1 )receptor agonist, or any other incretin mimetic 1 month prior to the planned study drug, or other drugs that the investigator believes may affect the trial;
* Those who took prescription or similar over-the-counter medications within 1 month prior to the trial to promote weight loss (eg, orlistat, sibutramine, rimonabant, phenylpropanolamine or chlorpheniramine) ;
* Alcohol intake is more than 21 units of alcohol per week (male) / 14 units of alcohol per week(female) (1 unit ≈ 360mL beer, or 45mL spirits with 40% alcohol content, or 150mL wine) 3 months prior to the screening.
* Regular consumption of caffeine more than 600 mg per day in the past 3 months (1 cup of coffee contains about 100 mg of caffeine, 1 cup of tea contains about 30 mg of caffeine, and 1 can of Coke contains about 20 mg of caffeine);
* Those who have taken caffeinated products or drugs within 48 hours prior to the study;
* Taken more than 5 cigarettes per day in the past 3 months;
* The investigator considers that the subject's diet has a big difference in the ratio to normal protein, carbohydrate, and fat intake (eg, vegetarian)person;
* There are symptoms such as dermatitis or skin abnormalities at the site of administration;
* Participated in other drug studies within 3 months prior to the planned study drug or the time of the last test drug was less than 3 months prior to screening for the trial; or attempted to participate in other drug trials during the study;
* Pregnancy, lactation or blood human chorionic gonadotropin(HCG) positive in pregnancy test;
* Drug abuse screening, alcohol breath test positive;
* Failure to ensure full participation in the trial;
* Others who have been judged by the investigator that inappropriate to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 28
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 0,0.25,1,4,6,8,12,24,36,48,60,72,96,144,192,264,336,648h
  Area under the plasma concentration versus time curve (AUC) after administration of of TG103
Peak Plasma Concentration (Cmax) | 0,0.25,1,4,6,8,12,24,36,48,60,72,96,144,192,264,336,648h
  Peak Plasma Concentration (Cmax) after administration of of TG103
Time to maximum plasma concentration（Tmax） | 0,0.25,1,4,6,8,12,24,36,48,60,72,96,144,192,264,336,648hours
  Time to maximum plasma concentration（Tmax）after administration of of TG103
Half time (t1/2) | 0,0.25,1,4,6,8,12,24,36,48,60,72,96,144,192,264,336,648hours
  The half time of TG103 after administration are calculated.
Apparent clearance (CL/F) | 0,0.25,1,4,6,8,12,24,36,48,60,72,96,144,192,264,336,648hours
  To assess the apparent clearance (CL/F) after administration of TG103
Fasting blood glucose | 1,2,3,4,5,7days
  Changes in Fasting blood glucose compared to baseline
2-hour postprandial blood glucose | 1,2,3,4,5,7days
  Changes in 2-hour postprandial blood glucose compared to baseline
fasting insulin | -1,3days
  Changes in fasting insulin compared to baseline
fasting glucagon | -1,3days
  Changes in fasting glucagon compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: jintong li, Principal Investigator — China-Japan Friendship Hospital; li chen, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin J, Cui G, Mi N, Wu W, Zhang X, Xiao C, Wang J, Qiu X, Han M, Li Z, Wang L, Lu T, Niu H, Wu Z, Li J. Safety, pharmacokinetics, and pharmacodynamics of TG103, a novel long-acting GLP-1/Fc fusion protein after a single ascending dose in Chinese healthy subjects. Eur J Pharm Sci. 2023 Jun 1;185:106448. doi: 10.1016/j.ejps.2023.106448. Epub 2023 Apr 14. PMID 37062422